CLINICAL TRIAL: NCT00712647
Title: Caret and Retinol Efficacy Trial: The Caret Coordinating Center
Brief Title: Carotene and Retinol Efficacy Trial
Acronym: CARET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Gary Goodman, MD, Fred Hutchinson Cancer Research Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FHCRC IR-4239A; U01CA063673 (NIH); 4239A (Other: FHCRC)
Record Dates: First submitted 2008-07-08; First posted 2008-07-10 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — beta Carotene; Vitamin A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Asbestos-exposed participants and heavy smokers
  Interventions: Drug: Beta Carotene and Retinol
- 2 (Placebo Comparator): Asbestos-exposed participants and heavy smokers
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Beta Carotene and Retinol — Pilot participants (ppts):
  Asbestos-Exposed--15 mg/day beta-carotene + 25,000 IU/day retinol Heavy Smokers--30 mg/day beta-carotene + 25,000 IU/day retinol
  Vanguard & Efficacy ppts:
  Asbestos-exposed AND heavy smokers--30 mg/day beta-carotene + 25,000 IU/day retinol
  Arms: 1
Other: Placebo — Two placebos, one each/day
  Arms: 2

SUMMARY:
The Carotene and Retinol Efficacy Trial (CARET) was a randomized, double-blind, placebo-controlled trial of the cancer prevention efficacy and safety of a daily combination of 30 mg of beta-carotene and 25,000 IU of retinyl palmitate in 18,314 persons at high risk for lung cancer. CARET began in 1985, and the intervention was halted in January 1996, 21 months ahead of schedule, with the twin conclusions for definitive evidence of no benefit and substantial evidence of a harmful effect of the intervention on both lung cancer incidence and total mortality. CARET continued to follow and collect endpoints on their participants through 2005. During the active intervention phase of CARET, serum, plasma, whole blood, and lung tissue specimens were collected on participants. These biospecimens make up the CARET Biorepository.

The CARET Biorepository is a valuable resource for population-based studies of the major human cancers. During CARET's twenty years of follow-up (1985-2005), we have received reports of 1,445 participants with lung cancer, 901 with prostate cancer, 433 with breast cancer, 334 with bladder cancer, 332 with colon cancer, and 1,429 with other cancers. CARET is one of the few trials that has prospectively collected serum, plasma, whole blood, blood spots (for DNA), and lung cancer tumor specimens, as well as smoking history and serial food frequency questionnaires (in some individuals for up to 12 years) in populations at high risk for lung cancer. This wealth of information in over 18,000 individuals makes the CARET Biorepository a special resource for cancer researchers.

ELIGIBILITY:
Inclusion Criteria:

* Asbestos-exposed men who were:

  * current smokers or quit within 15 years prior to enrollment
  * had first exposure to asbestos on the job at least 15 years prior to enrollment
  * had chest X-ray positive for changes compatible with asbestos exposure according to ILO criteria; or had been employed in a protocol-defined high-risk trade for at least 5 years, at least 10 years prior to enrollment.
* Heavy Smokers, men and women:

  * cigarette smoking history of 20+ pack-years
  * either current smokers or had quit within previous 6 years

Exclusion Criteria:

* Pre-menopausal women
* History or cirrhosis or hepatitis within 12 months prior to enrollment
* Taking > 5500 IU daily vitamin A supplement
* Taking any beta-carotene supplement
* History of cancer within 5 years prior to enrollment
* SGOT > than 2.5X upper limit of normal, or alkaline phosphatase > 1.5X upper limit of normal
* taking less than 50% of study vitamins during the enrollment period between the First and Second Visits.

Ages: 45 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18314 (Actual)
Dates: Start 1985-05; Primary Completion 2004-12 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Lung Cancer Incidence | bi-annual

SECONDARY OUTCOMES:
Other cancers | bi-annual

CONTACTS AND LOCATIONS:
Overall Officials: Gary E Goodman, MD, Principal Investigator — Fred Hutchinson Cancer Center